CLINICAL TRIAL: NCT00006209
Title: A Phase I Open-Label Dose Escalation Trial of Tucaresol in HIV-1 Infected Subjects Taking Potent Antiretroviral Therapy
Brief Title: A Study of Tucaresol in HIV-Infected Patients Who Are Taking Other Anti-HIV Drugs
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aaron Diamond AIDS Research Center (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 311A
Record Dates: First submitted 2000-09-11; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-06

CONDITIONS: HIV Infections
Keywords: HIV-1; Immunity, Cellular; Drug Therapy, Combination; CD4-Positive T-Lymphocytes; Antigens; Anti-HIV Agents; Viral Load; tucaresol
MeSH Terms: conditions — HIV Infections | interventions — tucaresol

INTERVENTIONS:
Drug: Tucaresol

SUMMARY:
The purpose of this study is to see if it is safe to give tucaresol to HIV-infected patients who are taking combination anti-HIV therapy (HAART). This study also examines the effect tucaresol has on viral load (level of HIV in the body) when tucaresol is used with HAART.

DETAILED DESCRIPTION:
Patients are enrolled sequentially into the next available dosage cohort. Each cohort receives a single dose of tucaresol, is observed for 2 weeks, and then receives 3 alternate-day doses of drug and careful safety monitoring, including 4 weeks follow-up after the final dose. Dose cohorts receive drug sequentially, the lowest-dose cohort receiving the drug first. Dose escalation may not proceed to the next higher-dose cohort until all patients from the prior lower-dose cohort have completed the 4-week follow-up after the multiple dosing, adverse events are within the described bounds, and the FDA has reviewed the safety information from the treated cohort and approved the dose escalation. The drug is administered 4 times within the 8 weeks of the study period. Weekly visits are required. Patients receive financial compensation.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are at least 18 years old.
* Are HIV-positive.
* Have more than 300 CD4 T cells/microL at screening.
* Are taking certain anti-HIV drugs.
* Have been taking these anti-HIV drugs successfully for at least 6 months.
* Do not expect to change their anti-HIV therapy while they are in the study.
* Have had plasma viral load less than 50 copies/ml while on their anti-HIV therapy.
* Have viral load that cannot be detected at screening and baseline tests.
* Are able to complete weekly visits.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Cannot give informed consent.
* Have abnormal laboratory test results at baseline.
* Are pregnant or breast-feeding.
* Have had certain short-term or long-term illnesses (such as heart disease, sickle cell disease, anemia, or lung problems).
* Have received a vaccination within the 30 days prior to enrollment.
* Have received any other experimental drug within 60 days of enrollment.
* Are taking abacavir (Ziagen, GW1592) or drugs that affect the immune system, such as IL-2, GM-CSF, corticosteroids, or cyclosporine.
* Have a history of tumors.
* Are actively using illegal drugs (methadone is allowed).
* Have hepatitis B or hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2000-06

CONTACTS AND LOCATIONS:
Locations (1):
- Rockefeller Univ, New York, New York, United States